CLINICAL TRIAL: NCT07193992
Title: Assessment of Non Vascular Risk Factors for Severity of Diabetic Foot Ulcers
Brief Title: Assessment of Non Vascular Risk Factors for Severity of Diabetic Foot Ulcers (DFUs)
Acronym: DFUs
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Essam Eldin Rshad Mohammed, Resident Physician, Department of Internal Medicine, Assiut University ., Assiut University
Other Study IDs: Diabetic foot ulcers
Record Dates: First submitted 2025-08-30; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcers; Diabetes Mellitus
Keywords: DFUs; Risk factors; Non vascular; Assessment; Diabetic foot ulcers; Amputation; Diabetes complications; Osteomyelitis; Glycemic control
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Diabetes Complications; Osteomyelitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes mellitus is a chronic disease that occurs either when pancreas does not produce enough insulin or when the body can't use it effectively. Diabetes mellitus include : type 1(insulin deficiency) , type 2 ( insulin resistance ) , gestational diabetes, maturity onset diabetes of the young ( MODY) , neonatal DM , wolfram syndrome, latent autoimmune diabetes in adults ( LADA ) , type 3 c diabetes, steroids - induced diabetes, cystic fibrosis disease ,Type 5 diabetes( Malnutrition related diabetes) which affect between 20-25 million primarily in Asia & Africa. According to WHO the number of living people with diabetes rose from 200 million in 1990 to 830 million in 2022 . According to IDF : The latest atlas 2025 report that 11.1% or 1- 9 of adult population ( 20 - 79 ) is living with diabetes, which 4 in 10 unaware of their condition. One of the serious complications is Diabetic foot ulcers . The global prevalence of DFU is around 6.3 % while the annual incidence reported between9.1 to 26.1 million cases, that's mean that 1 in 16 of diabetic patients experiences a DFUs . DFUs can be defined as wound or ulceration on the foot of diabetic patients due to a combination of factors such as neuropathy, peripheral artery disease, trauma or pressure . DFUs can lead to serious complications up to death like infection, osteomyelitis, limb amputation that significantly impact a person's quality of life, causing pain, disability and psychological distress. Beyond that immediate impact on patients, but also affect their families, and the healthcare system so it's considered as an economic burden due to health care costs and lost productivity. So to solve the problem we should know what cause it first and so we can prevent it before happening, not just finding a solution and that will affect not just the patients and their families, but also the country. Non vascular risk factors significantly impact DFU severity and healing including neuropathy, infection, poor glycemic control, obesity , inadequate foot care, certain immunological and inflammatory responses , age , malnutrition, smoking, High BMI , repetitive stress and pressure, certain foot conditions like onychomycosis and even iron deficiency anemia have been linked to it .

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic disease that arises either from insufficient insulin production by the pancreas or from the body's inability to use insulin effectively. It encompasses a wide spectrum of subtypes, including type 1 diabetes (absolute insulin deficiency), type 2 diabetes (insulin resistance), gestational diabetes, maturity-onset diabetes of the young (MODY), neonatal diabetes, Wolfram syndrome, latent autoimmune diabetes in adults (LADA), type 3C diabetes, steroid-induced diabetes, cystic fibrosis-related diabetes, and malnutrition-related diabetes, which affects approximately 20-25 million people primarily in Asia and Africa . According to the World Health Organization (WHO), the global number of people living with diabetes increased dramatically from 200 million in 1990 to 830 million in 2022 . The latest International Diabetes Federation (IDF) Atlas (2025) reports that 11.1% of adults aged 20-79 years-equivalent to one in nine-are living with diabetes, with nearly 40% of them unaware of their condition .

One of the most serious and costly complications of diabetes is the diabetic foot ulcer (DFU). Globally, the prevalence of DFUs is estimated at around 6.3%, with an annual incidence ranging from 9.1 to 26.1 million cases . This implies that roughly one in sixteen people with diabetes will experience a foot ulcer during their lifetime. DFUs are defined as wounds or ulcerations on the feet of individuals with diabetes, typically resulting from a combination of neuropathy, peripheral artery disease, trauma, and increased plantar pressure . These ulcers may progress to severe complications, including deep infection, osteomyelitis, and lower-limb amputation, leading not only to pain, disability, and psychological distress, but also to increased mortality . Beyond their devastating impact on patients and their families, DFUs pose a significant economic burden on healthcare systems due to high treatment costs and loss of productivity .

To reduce this burden, a clear understanding of the underlying risk factors is critical-not only to treat but also to prevent DFUs. In addition to vascular impairment, non-vascular risk factors have been shown to play a central role in ulcer development, severity, and healing. These include peripheral neuropathy, poor glycemic control, obesity, malnutrition, smoking, repetitive stress and pressure, inadequate foot care, infections such as onychomycosis or tinea pedis, high body mass index, and systemic conditions such as iron-deficiency anemia . Recent studies further emphasized the role of hematologic and nutritional abnormalities (e.g., anemia, hypoalbuminemia , elevated inflammatory markers) as independent predictors of ulcer severity . A systematic assessment of these non-vascular contributors enables clinicians to identify patients at higher risk, tailor treatment strategies, and implement preventive measures at earlier stages. When combined with vascular evaluation, this approach provides a comprehensive risk profile, improves clinical outcomes, reduces the need for amputation. and ultimately enhances quality of life for individuals with diabetes .

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 1 or type 2 diabetes mellitus
* Age ≥ 18 years
* Presence of diabetic foot ulcers (DFUs)
* Hemodynamically stable
* Willing and able to provide written informed consent prior to enrollment.

Exclusion Criteria:

* Diabetes complicated by peripheral vascular disease
* Non-diabetic foot ulcers, including venous ulcers or pressure ulcers
* Severe comorbid conditions (e.g., terminal illness or severe cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with Type 1 or Type 2 diabetes mellitus diagnosed with diabetic foot ulcers, recruited from Assiut University Hospitals. Patients with peripheral vascular disease, non-diabetic foot ulcers, or severe comorbidities will be excluded .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer recurrence rate | 1 year
  Title: Ulcer recurrence rate Description: Proportion of patients experiencing recurrence of diabetic foot ulcer during the study period, confirmed by clinical examination.
  Unit of Measure: Percentage of participants (%) Time Frame: 1 year

SECONDARY OUTCOMES:
1)Determine the modifiable non vascular risk factors . 2)Determine the severity & understanding the impact on healing , recurrence & outcomes. | 1 year
  Title: Wound size Description: Measurement of ulcer area (length × width) in cm² from baseline to study completion.
  Unit of Measure: cm²
  Title: Wound depth Description: Measurement of ulcer depth from the skin surface in centimeters. Unit of Measure: cm
  Title: Wound site Description: Anatomical location of the ulcer classified as forefoot, midfoot, or hindfoot.
  Unit of Measure: Site category
  Title: Wound characteristics Description: Assessment of wound features including skin integrity, presence of necrotic tissue, slough or eschar, exudate, and clinical signs of infection.
  Unit of Measure: Categorical assessment (presence/absence)
  Title: Ulcer severity using SINBAD classification Description: Assessment of ulcer severity using the SINBAD scoring system (Site, Ischemia, Neuropathy, Bacterial Infection, Area, Depth).
  Unit of Measure: Score (0-6).
Ulcer recurrence rate | 1 year
  Description: Proportion of patients experiencing ulcer recurrence during the study period.
  Unit of Measure: Percentage of participants (%)
1) Determine the modifiable non vascular risk factors (2) Determine the severity & understanding the impact on healing , recurrence & outcomes | 1 year
  Primary Outcome Measure:
  Title: Ulcer recurrence rate Description: Proportion of patients experiencing recurrence of diabetic foot ulcer during the study period, confirmed by clinical examination.
  Unit of Measure: Percentage of participants (%)
  Secondary Outcome Measures:
  Title: Wound size Description: Measurement of ulcer area (length × width) in cm² from baseline to study completion.
  Unit of Measure: cm² Unit of Measure: Site category Title: Wound characteristics Description: Assessment of wound features including loss of skin integrity, presence of necrotic tissue, slough or eschar, exudate or drainage, and clinical signs of infection.
  Unit of Measure: Categorical assessment (presence/absence). Title: Ulcer severity using SINBAD classification Description: Assessment of ulcer severity using the SINBAD scoring system (Site, Ischemia, Neuropathy, Bacterial Infection, Area, Depth).
  Unit of Measure: Score (0-6).

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mohammed Soliman, Professor, Study Chair — Assuit university - Endocrinology unit at internal medicine department.; Hanaa Mohammed Riad Hussien, Lecturer, Study Director — Assuit university - Endocrinology unit at internal medicine department.

IPD SHARING:
Plan to Share IPD: Undecided
All the study information l will share with others for increasing the general knowledge about the disease and aiming for adding something.